CLINICAL TRIAL: NCT02056587
Title: Everolimus (Afinitor) in Patients With Metastatic Renal Cell Carcinoma Following Progression on Prior Bevacizumab Treatment
Brief Title: Everolimus in Patients With Metastatic Renal Cell Carcinoma Following Progression on Prior Bevacizumab Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kidney Cancer Research Bureau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001LRU02T
Record Dates: First submitted 2014-02-04; First posted 2014-02-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: renal cell carcinoma; kidney cancer; bevacizumab failure; everolimus
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus (Experimental): All patients with metastatic renal cell carcinoma progressing on prior treatment with bevacizumab ± interferon enrolled into this study will receive everolimus in the dose of 10 mg daily until the disease progression or unacceptable toxicity.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — All patients with metastatic renal cell carcinoma progressing on prior treatment with bevacizumab ± interferon enrolled into this study will receive everolimus in the dose of 10 mg daily until the disease progression or unacceptable toxicity.

SUMMARY:
An estimated 10,000 metastatic renal cell carcinoma (RCC) patients receive first-line therapy in the Russian Federation. Bevacizumab (Avastin) in combination with interferon-alpha (IFN) is a recommended first-line treatment for metastatic RCC according to clinical recommendations of Russian Ministry of Health from 15.07.2010. Two randomized phase III trials (AVOREN, CALGB) showed that 50% of patients will progress on bevacizumab plus IFN within 8.5 - 10.2 months and will need sequential therapy.

Everolimus (Afinitor) is a single agent which was evaluated and demonstrated efficacy in randomized phase III study (RECORD-1) in metastatic RCC patients after failure of targeted therapy. However, in this trial everolimus was compared with placebo for the treatment of patients whose disease had progressed on treatment with sunitinib or sorafenib (n=227). Only 9% (n=24) of patients received bevacizumab. Thus, efficacy data of everolimus in patients with disease progression on first-line bevacizumab is limited.

Evaluating the effectiveness of everolimus in metastatic RCC patients with failure on bevacizumab with/without interferon alpha has a scientific and practical sense, and it is important for Russian Federation.

DETAILED DESCRIPTION:
17563 new cases of renal cancer and 83790 associated deaths have recorded in the Russian Federation in 2008. Renal cell carcinoma (RCC) is responsible for 4,3% of all malignancies, with increased risk of disease after the age of 60 years. Renal cell carcinoma accounts for 90% renal neoplasms, and in 85% of renal cell carcinoma cases light-cell morphology is diagnosed. Papillary, chromophobic cancer and cancer of the kidney collecting tubules.

30% patients with localized renal cell carcinoma are found to progress after surgical treatment. In the other 30% renal cell carcinoma is established at the dissemination stage. Therefore approximately 60% of renal cell carcinoma patients are estimated to have metastases.

According to estimations by Kidney Cancer Research Bureau, currently first line treatment is indicated to approximately 10,000 patients with metastatic renal cell carcinoma in Russia annually.

Until recently opportunities for systemic treatment in metastatic renal cell carcinoma were limited to administration of cytokines and clinical research investigating novel medications. Various combinations and doses of interleukin-2 (IL-2) and interferon-alpha (IFN) have been investigated in randomized studies in metastatic renal cell carcinoma. Immunotherapy was found to have only limited efficacy (overall response rate 15-16%, survival of 12 months). Therefore target medicines, specifically - tyrosine kinase inhibitors and mTOR inhibitors, are under development as first and subsequent lines of treatment.

According to standards of medical care established by the Ministry of Health and Social Development of the Russian Federation as of July 15, 2010, combination of bevacizumab (Avastin™) and interferon is recommended as first line treatment. According to two randomized phase III trials (AVOREN, CALGB) more than half of patients are expected to require further treatment for disease progression in 8,5-10,2 months. Everolimus (Afinitor) is the only medicine that has been investigated in a phase III multicenter study (RECORD-1) as second and subsequent lines of treatment for metastatic renal cell carcinoma resistant to targeted agents. However, most patients (n=277) had received sunitinib or sorafenib prior to enrolment; only some of them (24 patients (9%) had received bevacizumab. Therefore currently convincing evidence of everolimus efficacy after progression on prior treatment with bevacizumab or bevacizumab + IFN is lacking.

Hence it is deemed reasonable and practically relevant to investigate everolimus efficacy in patients with metastatic renal cell carcinoma previously treated on bevacizumab-containing regimens, in the Russian Federation.

Efficacy endpoints

Primary:

Primary endpoint is the proportion of progression-free patients for 2 months (based on results of a phase III study)

Secondary:

Median progression-free survival and overall survival from the time of enrolment Response rate, according to RECIST 1.1 Treatment safety and tolerability according to NCI-CTCAE v.4.0 Patients quality of life, according to EORTC QLQ-C30 questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven renal cell carcinoma
* CT-confirmed measurable disease
* Disease progression after bevacizumab +/- IFN
* Favorable/intermediate prognosis according to MSKCC
* Nephrectomy
* No contradictions to everolimus
* Age 18 or older
* Written informed consent

Exclusion criteria

* prior TKI's or mTOR inhibitor
* pregnant or nursing
* history of serious cardiac arrhythmia, congestive heart failure, angina pectoris, or other severe cardiovascular disease (i.e., New York Heart Association class III or IV)
* CNS metastases by neurologic exam and/or MRI
* local and/or systemic infections requiring antibiotics within 28 days prior to study entry
* other malignancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-11; Primary Completion 2013-04 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is the proportion of progression-free patients for 2 months (based on results of a phase III study) | 2 months

SECONDARY OUTCOMES:
Median progression-free survival | 12 months
Median overall survival | 24 months
Response rate according to RECIST 1.1 | 24 months
Treatment safety and tolerability according to NCI-CTCAE v.4.0 | 24 months

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Tatarstan Regional Cancer Center, Kazan', Tatarstan Republic
  - Altai Regional Cancer Center, Barnaul
  - N.N. Blokhin Russian Cancer Research Center, Moscow

REFERENCES:
- [Derived] Tsimafeyeu I, Snegovoy A, Varlamov S, Safina S, Varlamov I, Gurina L, Manzuk L. Everolimus in patients with metastatic renal cell carcinoma previously treated with bevacizumab: a prospective multicenter study CRAD001LRU02T. Target Oncol. 2015 Sep;10(3):423-7. doi: 10.1007/s11523-014-0347-4. Epub 2014 Dec 4. PMID 25466382